CLINICAL TRIAL: NCT00006079
Title: A Randomized Double-Blind Study of Alpha-Difluromethylornithine (DFMO) Versus Placebo in Patients With Cervical Intraepithelial Neoplasia (CIN) Grade 2-3
Brief Title: Eflornithine To Prevent Cervical Cancer in Patients With Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: ID92-026; P30CA016672 (NIH); MDA-ID-92026 (Other: UT MD Anderson Cancer Center); NCI-P00-0149; CDR0000067921 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-08-03; First posted 2004-05-26 (Estimated); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer; Precancerous Condition
Keywords: cervical cancer; cervical intraepithelial neoplasia grade 2; cervical intraepithelial neoplasia grade 3; Eflornithine
MeSH Terms: conditions — Uterine Cervical Neoplasms; Precancerous Conditions; Uterine Cervical Dysplasia | interventions — Eflornithine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm I (Experimental): Arm I-II: Patients receive one of two different doses of oral eflornithine daily. Treatment continues for 28 days.
  Interventions: Drug: Eflornithine
- Arm II (Experimental): Arm I-II: Patients receive one of two different doses of oral eflornithine daily. Treatment continues for 28 days.
  Interventions: Drug: Eflornithine
- Arm III (Placebo Comparator): Arm III: Patients receive oral placebo daily. Treatment continues for 28 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Eflornithine — Arm I-II: Patients receive one of two different doses of oral eflornithine daily for 28 days.
  Arms: Arm I; Arm II
Other: Placebo — Patients receive oral placebo daily for 28 days.
  Arms: Arm III

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. The use of eflornithine may be an effective way to prevent the recurrence of or further development of cervical cancer.

PURPOSE: Randomized phase II trial to determine the effectiveness of eflornithine in preventing cervical cancer in patients who have cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the efficacy of eflornithine versus placebo in causing regression in patients with cervical intraepithelial neoplasia. II. Compare the qualitative and quantitative toxicities of these treatment regimens in these patients. III. Establish the biochemical tissue markers of DNA content, PCNA, the ras oncogene, EGFR, and keratin and involucrin as intermediate biomarker end points for squamous carcinogenesis in these patients.

OUTLINE: This is a randomized, double blind, multicenter study. Patients are randomized to one of three treatment arms. Arm I-II: Patients receive one of two different doses of oral eflornithine daily. Arm III: Patients receive oral placebo daily. Treatment continues for 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed at 28 days, and then at 6, 12, 18, and 24 months.

PROJECTED ACCRUAL: A total of 180 patients (60 per treatment arm) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1) Women with newly diagnosed or recurrent CIN grade 2-3, involving an area 3times larger than the biopsy site. Patients must be > 18 years old, with a performance status less than or equal to 2 (Zubrod Scale) and a predicted life expectancy of greater than or equal to 12 months. Patients must have a medically safe form of contraception for the duration of the study. All patients must complete the of pretreatment evaluation, consent to colposcopy and cervical biopsy for histologic evaluation

Exclusion Criteria:

1) Patients may not have had a prior malignancy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 1998-06-19 (Actual); Primary Completion 2004-04-27 (Actual); Study Completion 2004-04-27 (Actual)

PRIMARY OUTCOMES:
Efficacy Comparison of Eflornithine versus Placebo | 28 Days
  Efficacy in causing regression in patients with cervical intraepithelial neoplasia measured by absence of disease progression or unacceptable toxicity. Patients are followed at 28 days, and then at 6, 12, 18, and 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Michele Follen, MD, PhD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- University of Texas - MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org